CLINICAL TRIAL: NCT00909220
Title: Translating Affective Science to Predict Outcomes of Behavioral Treatment for MDD
Brief Title: Using Affective Differences to Predict Response to Behavioral Treatment for Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Chicago (Other); Dartmouth College (Other)
Responsible Party: Principal Investigator, Jacqueline Gollan, Associate Professor of Psychiatry and Behavioral Sciences, Northwestern University
Other Study IDs: R21MH082133 (NIH); R21MH082133 (NIH)
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2018-01-16 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Depression
Keywords: Major Depressive Disorder, EEG, Negativity bias
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Current Major Depressive Disorder: Forty-one participants with a primary diagnosis of major depression using the Diagnostic and Statistical Manual of Mental Disorders (4th ed.; DSM-IV) and scores > 24 on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-C; Rush et al., 1986) were enrolled into a treatment study at Northwestern University's Feinberg School of Medicine in Chicago, Illinois. This group will receive Behavioral Activation psychotherapy.
  Interventions: Behavioral: Behavioral Activation
- Healthy Participants: Another 36 participants with no lifetime psychiatric symptoms and scores < 11 on the IDS-C were tracked prospectively, naturalistically, for 16 weeks.

INTERVENTIONS:
Behavioral: Behavioral Activation — Behavioral Activation included up to 16 weekly 50 minute psychotherapy sessions using BA (Addis & Martell, 2004; Martell et al., 2001, 2010). Techniques included functional analyses to identify the antecedent and consequential aspects of low mood, and interventions such as monitoring daily activities, assessing pleasure/satisfaction and competence achieved via activities, assigning tasks that induce mastery or pleasure, and reducing skill deficits. Clinicians included postdoctoral fellows in clinical psychology (n = 2) or licensed clinical psychologists (n = 2).
  Groups: Current Major Depressive Disorder

SUMMARY:
This study will determine how people with depression differ from healthy people in brain activity and interpreting emotions, both before and after receiving a psychotherapy treatment.

DETAILED DESCRIPTION:
Major depressive disorder is a serious form of depression that may be treated with psychotherapy. However, up to 40% of adults with depression do not show reduced symptoms when treated with cognitive therapy or behavioral activation (BA), two common forms of psychotherapy. Certain indicators are generally linked with a successful outcome of psychotherapy-demographic and clinical characteristics, comorbidity, and treatment adherence-but no factors reliably predict outcomes of psychotherapy in individuals. This study will test whether two characteristics related to the way people process emotions, affective asymmetry and affective reactivity, can predict whether people with depression will improve with BA therapy.

Both depressed and healthy participants will be recruited for this study. Participation in this study will last 31 weeks. All participants will complete baseline assessments at Weeks 1 and 2. Depressed participants will then begin receiving 16 weekly sessions of BA therapy. All participants will be assessed again after 8, 16, 17, and 28 weeks. Assessments will include the following: a urine toxicology screening; interviews on mental and physical health, family and childhood experiences, and current mood and functioning; computer tasks; recordings of electroencephalography (EEG) activity; recordings of reaction to a startle probe; recordings of electromyography (EMG) activity; recordings of electrodermal activity (EDA); and measurement of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants should have no lifetime history of psychiatric disorder
* Depressed participants should have a current diagnosis of major depressive disorder, as defined by the DSM-IV

Exclusion Criteria:

* History of bipolar affective disorder
* History of psychosis
* Current non-psychotic Axis I disorder, if it constitutes the predominant aspect of the clinical presentation and immediately requires treatment other than that offered in the study
* History of substance dependence within the past 6 months
* Antisocial, borderline, schizotypal, or schizoid personality disorders
* Evidence of any medical disorder or condition that could cause depression or preclude the use of study treatments
* Current treatment with catecholaminergic antihypertensive medication, such as reserpine, beta-blockers, clonidine, and alphamethyldopa
* Current use of antidepressant medication
* Clear indication of secondary gain
* Current suicide risk sufficient to preclude treatment on an outpatient basis
* Severe, unstable concurrent psychiatric conditions likely to require hospitalization within 6 months of study entry
* Already receiving a targeted psychotherapy aimed at depression

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are drawn from the general population through on-line advertisements for the study.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline K. Gollan, PhD, Principal Investigator — Northwestern University

IPD SHARING:
Plan to Share IPD: Yes
Request PI (JGollan) for de-identified data at j-gollan@northwestern.edu
Supporting Information: Study Protocol, SAP
Time Frame: 01/01/18-01/01/20
Access Criteria: 01/01/18-01/01/20

REFERENCES:
- [Result] Gollan JK, Hoxha D, Chihade D, Pflieger ME, Rosebrock L, Cacioppo J. Frontal alpha EEG asymmetry before and after behavioral activation treatment for depression. Biol Psychol. 2014 May;99:198-208. doi: 10.1016/j.biopsycho.2014.03.003. Epub 2014 Mar 24. PMID 24674708
- [Result] Gollan JK, Hoxha D, Hunnicutt-Ferguson K, Norris CJ, Rosebrock L, Sankin L, Cacioppo J. Twice the negativity bias and half the positivity offset: Evaluative responses to emotional information in depression. J Behav Ther Exp Psychiatry. 2016 Sep;52:166-170. doi: 10.1016/j.jbtep.2015.09.005. Epub 2015 Sep 26. PMID 26434794
- [Result] Gollan JK, Hoxha D, Hunnicutt-Ferguson K, Norris CJ, Rosebrock L, Sankin L, Cacioppo J. The negativity bias predicts response rate to Behavioral Activation for depression. J Behav Ther Exp Psychiatry. 2016 Sep;52:171-178. doi: 10.1016/j.jbtep.2015.09.011. Epub 2015 Sep 28. PMID 26433700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from each group were recruited from the same community locations via advertisements and the internet. Enrollment began 5/2009 and ended 7/2011.
Pre-assignment Details: All depressed participants were enrolled into the Behavioral Activation Treatment arm. All healthy participants were tracked for the duration of the study.
Groups:
- Current Major Depressive Disorder: Forty-one participants with a primary diagnosis of major depression using the Diagnostic and Statistical Manual of Mental Disorders (4th ed.; DSM-IV) and scores > 24 on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-C; Rush et al., 1986) were enrolled into a treatment study at Northwestern University's Feinberg School of Medicine in Chicago, Illinois.
  Behavioral Activation: 16 weekly study visits aimed at identifying avoidance patterns used in social or physical situations that contribute to depression and replacing them with reinforcing experiences using directive behavioral strategies
- Healthy Participants: Another 36 participants with no lifetime psychiatric symptoms and scores < 11 on the IDS-C were enrolled for assessment over 16 weeks
Period: Overall Study
Arm/Group | Current Major Depressive Disorder | Healthy Participants
Started | 41 (Started enrolling participants May 2009) | 36 (Started enrolling participants May 2009)
Data Entry | 41 | 36
Data Analyses | 41 | 36
Submission for Publication | 41 | 36
Completed | 41 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Current Major Depressive Disorder: participants with a primary diagnosis of major depression using the Diagnostic and Statistical Manual of Mental Disorders (4th ed.; DSM-IV) and scores > 24 on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-C; Rush et al., 1986).
  Additional inclusion criteria specified that participants should be between ages 18 and 65 years, medically healthy, medication-free, and with no medication washout. Exclusion criteria included lifetime bipolar disorder, psychosis, obsessive-compulsive disorder, substance abuse/dependence, and several personality disorders (i.e., borderline, schizoid, schizotypal, antisocial).
  Behavioral Activation: 16 weekly study visits aimed at identifying avoidance patterns used in social or physical situations that contribute to depression and replacing them with reinforcing experiences using directive behavioral strategies.
- Healthy Participants: participants with no lifetime psychiatric symptoms and scores < 11 on the IDS-C were enrolled for assessment over 16 weeks. Additional inclusion criteria specified that participants should be between ages 18 and 65 years, medically healthy, medication-free, and with no medication washout. Exclusion criteria included lifetime bipolar disorder, psychosis, obsessive-compulsive disorder, substance abuse/dependence, and several personality disorders (i.e., borderline, schizoid, schizotypal, antisocial).).
- Total: Total of all reporting groups
Arm/Group | Current Major Depressive Disorder | Healthy Participants | Total
Number analyzed (Participants) | 41 | 36 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 36 | 77
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (12) | 35 (14) | 35 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 20 | 46
  Male | 15 | 16 | 31
Region of Enrollment [Number; unit: participants]
  United States | 41 | 36 | 77

OUTCOME MEASURES:

1. Primary Outcome: Analyses of Covariance to Test for Group Differences (MDD vs. Healthy) on Clinician-rated Depression Severity After 16 Weeks of Behavioral Activation Psychotherapy, Controlling for Baseline Depression Severity.
Description: The Inventory of Depressive Symptomatology-Clinician Rated measure (IDS-C; Rush, Giles, Schlesser, Fulton, Weissenburger, Burns, 1986; Rush, Carmody, & Reimitz, 2000; Rush, Trivedi, Ibrahim, Carmody, Arnow, Klein, et al., 2003) is a 30-item measure that reflects the presence and severity of DSM-IV symptoms of depression. The item scores on this scale are summed to create a total score. Scores range from 0 (minimum score, reflecting no symptoms) to 84 (maximum score, reflecting highest severity). Scores between 0-11 are interpreted as 'no depression'; scores between 12-23 are interpreted as 'mild severity'; scores between 24-36 are interpreted as 'severe'; and total scores between '47-84' are interpreted as 'very severe'.
Time Frame: Week 16
Population: Intent to treat sample.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Current Major Depressive Disorder: Forty-one participants with a primary diagnosis of major depression using the Diagnostic and Statistical Manual of Mental Disorders (4th ed.; APA. DSM-IV) and scores > 24 on the Inventory of Depressive Symptomatology-Clinician Rated (IDS-C; Rush et al., 1986).
- Healthy Participants: An additional 36 participants with no lifetime psychiatric symptoms and scores < 11 on the IDS-C were enrolled
Arm/Group | Current Major Depressive Disorder | Healthy Participants
Number analyzed (Participants) | 41 | 36
units on a scale | 14.1 (10.1) | 2.7 (2.7)
Statistical Analysis 1: Comparison: Current Major Depressive Disorder vs Healthy Participants; ANCOVA comparing groups (HEA v MDD), controlling for baseline depression (IDS-C score at week 0) to estimate depression at the end of treatment (IDS-C score at week 16); Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.27 to 0.49], Standard Error of Mean 0.06

2. Primary Outcome: Analyses of Covariance to Test for Group Differences (MDD vs. Healthy) on Patient-rated Depression Severity After 16 Weeks of Behavioral Activation Psychotherapy, Controlling for Baseline Depression Severity.
Description: The Inventory of Depressive Symptomatology, Self-Rated measure (IDS-SR; Rush et al., 1986, 2003) is a 30-item measure of depression severity completed by the participant. The item scores on this scale are summed to create a total score (range from 0 (no symptoms) to 84 (highest severity). The item scores on this scale are summed to create a total score (range from 0 (minimum score reflecting no symptoms) to 84 (maximum score, reflecting highest severity). Severity of depression is reflected by total score (e.g., scores between 0-13 is interpreted as 'no depression', scores between 14-25 are interpreted as 'mild severity'; total scores between 26-48 are interpreted as 'severe', and total scores between '49-84' are interpreted as 'very severe'.
Time Frame: Week 16
Population: Intent to treat sample.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Current Major Depressive Disorder | Healthy Participants
Number analyzed (Participants) | 41 | 36
units on a scale | 16.9 (13.4) | 3.0 (4.6)
Statistical Analysis 1: Comparison: Current Major Depressive Disorder vs Healthy Participants; ANCOVA comparing groups (HEA v MDD), controlling for baseline depression (IDS-SR score at week 0) to estimate depression at the end of treatment (IDS-SR score at week 16); Test type: Superiority — ANCOVA; p < 0.05, ANCOVA; Mean Difference (Final Values) = 0.39, 95% CI 2-sided [0.31 to 0.59], Standard Error of Mean 0.07

3. Primary Outcome: Pre-treatment Frontal EEG Asymmetry Score as a Predictor of Negative Affect at Post-treatment
Description: Frontal EEG asymmetry scores were calculated over the midfrontal sites, subtracting the natural log of the alpha power of the electrode in the left hemisphere (F3 or F7) from that of the right frontal electrode (F4 or F8), creating one summary alpha asymmetry variable. The absolute value of this difference score was taken. Using the natural log transformation is used in EEG asymmetry research as EEG power appears to be positively skewed. A higher score thus reflected greater relative left versus right frontal activation (e.g., relatively higher right alpha activity).
Time Frame: Week 0
Measure: Mean (Standard Error); unit: Alpha power
Groups:
- Current Major Depressive Disorder: participants diagnosed with current major depressive disorder per the Structured Clinical Interview for the DSM-IV Axis I Disorders, (SCID; First, Spitzer, Gibbon, & Williams, 2002) and a score > 24 on the Inventory of Depressive Symptomatology-Clinician-Rated, (IDS-C; Rush et al., 2003; Rush et al., 1986).
- Healthy Participants: Healthy participants were enrolled with no lifetime history or current presentation of psychiatric symptoms per the SCID and a score < 11 on the IDS-C.
Arm/Group | Current Major Depressive Disorder | Healthy Participants
Number analyzed (Participants) | 37 | 35
Alpha power | 0.43 (0.12) | 0.16 (0.05)
Statistical Analysis 1: Comparison: Current Major Depressive Disorder vs Healthy Participants; Test type: Other — Multiple regression analyses; p = .02, Regression, Linear — p <0.05 a priori threshold for statistical significance; beta = 0.43, Standard Error of Mean 6.75

4. Primary Outcome: A Two Level Hierarchical Model Testing the Association Between Negativity Bias Change During BA Treatment With Patient-reported Depression Severity (Week 16 IDS-SR).
Description: The negativity bias, characterized as the tendency to evaluate unpleasant versus pleasant information as more important, was measured using a computer task. Sitting in front of the computer, participants viewed emotionally evocative images and assigned their evaluations of how the intensity of these emotional images using a grid. The grid is comprised of a matrix, with 5 points on the horizontal axis representing the positivity seen in the image (0=not at all, 4 = extremely positive) by 5 points on a vertical axis representing the negativity seen in the image (0=not at all, 4 = extremely negative) matrix. The dimensional variable, negativity bias, is calculated as the difference in the mean ratings of very unpleasant images minutes the positive ratings of the very pleasant images. The Inventory of Depressive Symptomatology, Self-Rated (IDS-SR; Rush et al., 1986, 2003) is a 30-item measure of depression severity provided by the participant.
Time Frame: Weeks 0-16
Population: First level units were 'weeks in BA treatment', with participants limited to those diagnosed with MDD and who attended five or more therapy sessions, resulting in a total of 421 treatment weeks for analysis. Second-level units were the 'MDD subjects entering treatment' (n = 41)
Measure: Geometric Least Squares Mean (Standard Error); unit: slope
Arm/Group | Current Major Depressive Disorder
Number analyzed (Participants) | 41
slope | -3.43 (0.75)
Statistical Analysis 1: Comparison: Current Major Depressive Disorder; A two-level hierarchical linear model assessing the effects of negativity bias and positivity offset at pre-treatment on the rate of depression severity (IDS-SR) over 16 weeks of treatment (time). First level units were 'weeks in BA treatment', with participants limited to those who attended five or more therapy sessions, resulting in a total of 421 treatment weeks for analysis. Second-level units were the 'subjects entering BA treatment'; Test type: Other — Hierarchical linear modeling (HLM) , an ordinary least square (OLS) regression-based analysis; p < 0.05, Regression, Logistic — The variation of slopes among participants for each variable were calculated. If significant, a second level of analysis focused on predictors of the variation was conducted; df = 31; Slope = 2.58, 95% CI 2-sided [1.22 to 2.77], Standard Error of Mean 0.75

ADVERSE EVENTS:
Time Frame: Serious and Other (Not including Serious) Adverse Events were not collected/assessed.
Groups:
- Current Major Depressive Disorder: Diagnosed with current major depressive disorder per the Structured Clinical Interview for the DSM-IV Axis I Disorders, (SCID) and a score ≥ 24 on the Inventory of Depressive Symptomatology-Clinician-Rated, (IDS-C).
- Healthy Participants: No lifetime history or current presentation of psychiatric symptoms per the SCID and a score ≤ 11 on the IDS-C.
Arm/Group | Current Major Depressive Disorder | Healthy Participants
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
We enrolled adults who were medication-free, which may limit the generalizability of these results to those individuals who rely on pharmacotherapy and somatic therapies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No